CLINICAL TRIAL: NCT03353259
Title: Tocilizumab (RoActemra) and Tranexamic Acid (Cyklokapron) Used as Adjuncts to Chronic Subdural Hematoma Surgery
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DMC concluded that the results of 382 included patients were clear.
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Milo Stanisic, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1512/REK nord; 2017-001670-42 (EudraCT Number)
Record Dates: First submitted 2017-10-17; First posted 2017-11-27 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Chronic Subdural Hematoma
MeSH Terms: conditions — Hematoma, Subdural, Chronic | interventions — Tranexamic Acid; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SS-TG (No Intervention): Standard surgery using burr-hole procedure, irrigation and drainage.
- SS-TXA-TG (Active Comparator): Standard surgery using burr-hole procedure, irrigation and drainage combined withTranexamic acid (Cyklokapron) administration. Cyklokapron tablets will be administered postoperatively in dosage 500 mg twice a day until complete hematoma disappearance.
  Interventions: Combination Product: Tranexamic acid and Tocilizumab
- SS-TXA-RoA (Active Comparator): Standard surgery using burr-hole procedure, irrigation and drainage combined with Tranexamic acid (Cyklokapron) and Tocilizumab (RoActemra) administration. Cyklokapron tablets will be administered postoperatively in dosage 500 mg twice a day combined with RoActemra subcutaneous injection of 162 mg once a week until complete hematoma disappearance.
  Interventions: Combination Product: Tranexamic acid and Tocilizumab

INTERVENTIONS:
Combination Product: Tranexamic acid and Tocilizumab — The first intervention is Tranexamic acid, The second intervention is Tocilizumab
  Other Names: Cyklokapron and RoActemra
  Arms: SS-TXA-RoA; SS-TXA-TG

SUMMARY:
Primary objectives of the study are to investigate whether adjuvant treatment in the form of Tranexamic acid (Cyklokapron) and Tocilizumab (RoAcmera) to surgery in patients with chronic subdural hematomaina can:

1. effectively decrease the rate of lesion recurrence requiring re-operation,
2. effectively shorten the time of lesion resolution.

Secondary objectives of the study are:1) assess the postoperative functional outcome and quality of life of participants, 2) assess the postoperative mortality of participants, 3) assess the treatment safety data, 4) assess the cure rate of participants.

DETAILED DESCRIPTION:
Primary endpoints in the study are: 1) determine postoperative recurrence requiring reoperation using clinical examination and CT imaging, 2) determine the time period necessary to complete healing using clinical examination and CT imaging.

Secondary endpoints in the study are: 1) to determine the functional outcome and quality of life of the participants using questionnaires, 2) to determine the mortality of the participants related to chronic subdural hematoma, 3) to determine the treatments complications and adverse events of the participants, 4) to determine the curation using clinical examination and CT imaging.

ELIGIBILITY:
Inclusion Criteria:

* patients with informed consent, without presenting of any known contraindication for the use of Tranexamic acid and Tocilizumab.

Exclusion Criteria:

* patients or relatives who refused to consent, presenting of any known contraindication for the use of Tranexamic acid and Tocilizumab.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Tocilizumab (RoActemra) and Tranexamic acid (Cyklokapron) used as Adjuncts to Chronic Subdural Hematoma Surgery Regarding Postoperative Recurrence | 6 months period after the initial surgery.
  To determine the rate in number and percentage of postoperative recurrence requiring re-operation

CONTACTS AND LOCATIONS:
Overall Officials: Milo Stanisic, Principal Investigator — Oslo University Hospital
Locations (1):
- Milo Stanisic, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No